CLINICAL TRIAL: NCT06286124
Title: Midline Restoration After HYbriD Incisional Hernia RepAir (HYDRA) With the SymbotexTM Mesh
Brief Title: Midline Restoration After HYbriD Hernia RepAir Surgery (HYDRA)
Acronym: HYDRA
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medtronic (Industry); Alrijne Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. Pieter J Tanis, Prof. dr., Erasmus Medical Center
Other Study IDs: 8612
Record Dates: First submitted 2023-12-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Incisional Hernia of Midline of Abdomen
Keywords: Incisional Hernia; Repair; Hybrid
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Incisional Hernia patients: Patients with an Incisional Hernia, who present in the participating center
  Interventions: Procedure: Hybrid Surgery

INTERVENTIONS:
Procedure: Hybrid Surgery — Hybrid incisional hernia repair, as described by Van den Dop et al. (2021)
  Other Names: three-step incisional hybrid repair (TIHR)

SUMMARY:
The goal of this observational study is to learn about the functioning of the abdominal wall in patients who underwent hybrid (open- and laparoscopic) incisional hernia repair. The main objective is to assess the anatomical restoration and function of the linea alba one year after surgery by ultrasonography and mean peak torque during trunk flexion using a BioDex machine.

DETAILED DESCRIPTION:
Rationale: Abdominal wall functioning has been reported to be higher in patients that underwent open incisional hernia repair compared to laparoscopic incisional hernia repair. With the use of a recently developed hybrid approach, we aim for a functional anatomical restoration of the linea alba while also achieving the technical advantages of the hybrid approach.

Objective: The main objective is to asses functional anatomical restoration of the linea alba through functioning in mean peak torque, and ultrasound examination.

Study design: Multicentre prospective cohort study. Study population: Adult patients with a midline incisional hernia ≥4 cm and ≤10 cm.

Intervention: Not applicable. Main study parameters/endpoints: The primary objective of this study is to assess anatomical restoration and function of the linea alba one year after surgery by ultrasonography and measuring the mean peak torque during trunk flexion using a BioDex(trademark) machine.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No risk is associated with participation other than known complications for incisional hernia repair. HYDRA is part of standard care in the Alrijne Hospital, and the technique has previously been published. The mesh used in this study is being used on a world-wide scale. We do not expect additional risks with this study. As participants have to visit the Erasmus Medical Center (Erasmus MC) an additional three times and have to fill in additional questionnaires, there is a burden for enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Scheduled for elective HYDRA-surgery
* Midline incisional hernia larger than 4 centimetres in mean width
* Sufficient knowledge of the Dutch language to be able to understand and fill in the questionnaires
* Signed informed consent form by patient

Exclusion Criteria:

* Pregnant at inclusion
* Inclusion in other trials with interference of the primary and secondary endpoints
* American Society of Anesthesiologists Classification (ASA Classification) > 3
* Hernia defect larger than 10 centimetres in mean width
* Incarcerated hernias or emergency procedure
* Unable to perform a trunk flexion
* Incapacitated patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for Hybrid repair of their incisional hernia
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Mean peak torque 1 year | 12 months
  The functioning of the abdominal wall in Nm/kg as assessed by a BioDex

SECONDARY OUTCOMES:
Mean peak torque 2 years | 24 months
  The functioning of the abdominal wall in Nm/kg as assessed by a BioDex
Recurrent Incisional Hernia | 1 month, 12 months and 24 months
  Ultrasonography examination of the abdominal wall for the detection of a recurrent incisional hernia.
Severity of surgical complications | 1 month
  Through Clavien-Dindo classification
Surgical complications | 1 month
  Type of complication will be recorded as a free-text field
General Quality of Life | pre-operative, 12 months and 24 months
  Measure quality of life using the Short Form Health Survey, a 36-question questionnaire
Mesh specific Quality of Life | 1 month, 12 months and 24 months
  The Carolina Comfort Scale, which is a mesh-specific quality of life questionnaire, will be used in order to assess satisfaction with the placed mesh.
Scar satisfaction | pre-operative, 1 day, 1 month
  Visual Analogue Scale for the how satisfied patients are with the new scar from the surgery, reaching from 0 to 10.
Pain in the abdominal region | pre-operative, 1 day, 1 month
  Visual Analogue Scale for pain in the region of the hernia reaching from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Tanis, Prof. dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Alrijne Hospital, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data is partly retrieved from patient files and from questionnaires (after informed consent). Even though the data is pseudonymized, there is too much risk of confidentiality breach.

REFERENCES:
- [Background] van den Dop LM, de Smet GHJ, Bus MPA, Lange JF, Koch SMP, Hueting WE. A new three-step hybrid approach is a safe procedure for incisional hernia: early experiences with a single centre retrospective cohort. Hernia. 2021 Dec;25(6):1693-1701. doi: 10.1007/s10029-020-02300-9. Epub 2020 Sep 12. PMID 32920734